CLINICAL TRIAL: NCT04779021
Title: Caracterisation of SARS-Cov2 Infected Patients Hospitalized in Infectious Disease Department
Brief Title: Caracterisation of COVID-19 Patients Hospitalized in Infectious Disease Department
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21infectiocovid01
Record Dates: First submitted 2021-02-23; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Covid19; SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Hospitalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Other: Hospitalisation for SARS-COV2 infection — Patients hospitalized for SARS-COV2 infection

SUMMARY:
The main objective of this cohort is to characterize COVID-19 patients hospitalized in infectious disease department. The collection of clinical and biological data from start of hospitalization to long-term follow up will contribute to a better description of the patient care, to the identification of predisposition to complication related to the disease, and to the evaluation of the impact of different therapeutical strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = to 18
* Patients hospitalised for SARS-CoV-2 infection confirmed by RT PCRand/or CT scan and/or serology

Exclusion Criteria:

* Patients for whom SARS-CoV-2 infection has not been confirmed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for SARS-COV2 infection
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical characteristics | 34 months
  Describe the clinical characteristic of patients hospitalized for SARS-CoV- 2 infection Identify factors associated with the COVID-19 disease severity
Biological characteristics | 34 months
  Describe the biological characteristic of patients hospitalized for SARS-CoV- 2 infection Identify factors associated with the COVID-19 disease severity
Radiological characteristics | 34 months
  Describe the radiological characteristic of patients hospitalized for SARS-CoV- 2 infection Identify factors associated with the COVID-19 disease severity

SECONDARY OUTCOMES:
Number of patient hospitalised for Covid-19 | 34 months
  Inpatient up to Day 28 or discharge
Overall Inpatient Mortality | 34 months
  Number of death due to Covid-19
Requirement for mechanical ventilation | 34 months
  Number of patients requiring mechanical ventilation
ICU Length of Stay (LOS) | 34 months
  Duration measured in days
Evolution of patient general state during hospitalisation | 34 months
  the different measures (Body Mass Index (BMI), respiratory rate at rest, peripheral oxygen saturation, need for oxygen supplementation, body temperature) will be aggregated in order to obtain a clinical status corresponding to the clinical evolution (good or bad) of the patient's general state.
Biological tests | 34 months
  Dosage of Lymphocytes, C-reactive protein and IL-6

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de NICE - Infectiologie, Nice
  - CHU de NICE - Urgences, Nice

IPD SHARING:
Plan to Share IPD: No
No data sharing plan is scheduled